CLINICAL TRIAL: NCT04007718
Title: Learning Effective New Strategies - Parkinson's Disease
Brief Title: Learning Effective New Strategies for Worry in Parkinson's Disease
Acronym: LENS-PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Lonneke van_Tuijl, Research associate, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HR-18/19-8816
Record Dates: First submitted 2019-06-24; First posted 2019-07-05 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease; Anxiety
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Behavioral: Interpretation bias training
- Control (Sham Comparator)
  Interventions: Behavioral: Interpretation bias training

INTERVENTIONS:
Behavioral: Interpretation bias training — Active: 50% positive endings to scenarios, 50% generation of positive endings to ambiguous scenarios Control: 100% ambiguous endings to scenarios with no instructions to imagine positive endings

SUMMARY:
High rates of anxiety and worry has been observed in people with Parkinson's (PwP). Previous research outside of PwP has shown that individuals with anxiety have a habit of interpreting ambiguous information in a negative manner (i.e., interpretation bias), and that it is possible to encourage a more positive interpretation bias through an online training.

In the current study, the aim is to test the acceptability and feasibility of an online training program that aims to encourage more positive interpretation bias in high worrying PwP. Participants complete an online baseline assessment, and are then invited to complete ten training sessions over a period of three weeks followed by another assessment and follow-up assessments (at 1 month & 3 months). Participants are randomized into either the active condition or control condition. Across both conditions, participants will listen to short, everyday scenarios which are ambiguous (could end positively or negatively). In the active condition, a positive ending is given in half of the scenarios. In the other half, participants are instructed to imagine positive endings to ambiguous scenarios. In the control condition, all scenarios end ambiguously and no instructions are given about imagining positive endings.

The primary aim of the study is to test the acceptability and feasibility of the online training platform. Participants will complete a feasibility interview after completing the training. Specifically, the acceptability of the following will be tested: i) the online nature of the training (and lack of face-to-face contact); ii) being randomised into one of the two conditions; iii) the number and duration of the assignments; and iv) the text messages/e-mail/phone call reminders to complete the assignments. The feasibility of the online training platform will be judged on the i) rate of recruitment; ii) retention rates during the training; iii) adherence to the study (i.e., number of assignments completed); iv) retention rates at follow-up. The secondary aim is to estimate the effect size of the active condition (vs. control; on worry scores post-training, and at follow-ups) to inform power analyses for a future randomised control trial.

It is hypothesised that the training will be acceptable and feasible in a high worrying PwP sample. It is also hypothesised that the training will be effective in reducing worry and improving interpretation bias.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's Disease
* can use a computer independently
* have (correct to) normal hearing
* scores above 62 on the Penn State Worry Questionnaire

Exclusion Criteria:

* Those who have previously taken part in lab-based studies at King's College London where measures of interpretation bias were included.
* Currently or have recently (past six months) received psychological treatment.
* If participants are currently taking anti-depressants or anti-anxiety medication, they need to have been stable on the same dose for at least six weeks.
* Participants who score 2 or higher on the ninth item of the Patient Health Questionnaire-- (measuring suicidal ideation) at screening will be excluded.
* If individuals do not have regular access to a computer and/or the internet, they will be excluded.
* Those who can not concentrated on the questions asked during the Modified Telephone Interview for Cognitive Status, or are confused by the questions asked.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability; rating of online training | At approximately 4 weeks (during the feasibility interview)
  Whether participants accept the online nature of the training (extent of positive feedback compared to negative feedback)
Acceptability; lack of face-to-face contact | At approximately 4 weeks (during the feasibility interview)
  Whether participants accept the lack of face-to-face contact
Acceptability; number of assignments | At approximately 4 weeks (during the feasibility interview)
  Whether participants accept the number of assignments
Acceptability; duration of assignments | At approximately 4 weeks (during the feasibility interview)
  Whether participants accept the duration of assignments
Acceptability; reminders | At approximately 4 weeks (during the feasibility interview)
  Whether participants accept the text messages/e-mail/phone call reminders
Acceptability; randomisation | Participants are asked during the eligibility call prior to starting the training if they are happy to be randomised. As such, acceptability to be randomised is at baseline.
  Proportion of eligible participants who agree to being randomised to those who do not agree
Training feasibility; rate of recruitment | From recruitment start (moment when Parkinson's UK [United Kingdom] advertise the study) till study close (either end of November, 2019, or when the recruitment target is met; approximately 5 months)
  The feasibility of the training based on the rate of recruitment
Training feasibility; retention rates | Duration of study (approximately 5 months)
  The feasibility of the training based on the retention rates during the training
Training feasibility; study adherence | Assignments are completed over three weeks, with a possibility of a one week extension for those who have not completed at least 8 in the three weeks.
  The feasibility of the training based on the adherence to the study (number of assignments completed)
Training feasibility; retention at one-month follow-up | Duration of study (approximately 5 months)
  The feasibility of the training based on the retention rates at follow-up (i.e., number of missing cases or drop outs at the one month follow-up)
Training feasibility; retention at three-month follow-up | Duration of study (approximately 5 months)
  The feasibility of the training based on the retention rates at follow-up (i.e., number of missing cases or drop outs at the three month follow-up)

SECONDARY OUTCOMES:
Decrease in worry (estimation of effect size); post-training | Baseline worry scores will be compared to worry scores after the training (assessment 2; completed approximately 3 weeks later)
  The extent that worry has changed from before to after training in the active condition compared to the control condition based on the Penn State Worry Questionnaire (scores can range from 16 to 80; higher scores indicate more worry)
Decrease in worry (estimation of effect size); at one-month follow-up | Baseline worry scores will be compared to worry scores at the one-month follow-up
  The extent that worry has changed from before training to the one month follow-up in the active compared to the control condition, as mediated by post-training worry scores, based on the Penn State Worry Questionnaire (scores can range from 16 to 80; higher scores indicate more worry)
Decrease in worry (estimation of effect size); at three-months follow-up | Baseline worry scores will be compared to worry scores at the three-months follow-up
  The extent that worry has changed from before training to three months after training in the active condition compared to the control condition, as mediated by post-training worry scores, based on the Penn State Worry Questionnaire (scores can range from 16 to 80; higher scores indicate more worry)

OTHER OUTCOMES:
Improvement in interpretation bias (scrambled sentences task) | Comparing baseline scores to post-training (assessment 2; completed approximately 3 weeks later) scores
  Whether scores on the scrambled sentences task have changed specifically in the training condition. The scrambled sentences tasks involves unscrambling 20 sentences to form either position or negative solutions and is calculated by the proportion of negative solutions to positive solution (i.e., higher scores = more negative interpretation bias).
Improvement in interpretation bias (recognition test) | Comparing baseline scores to post-training (assessment 2; completed approximately 3 weeks later) scores
  Whether scores on the recognition test have changed specifically in the training condition. The recognition test involves reading ten (ambiguous) scenarios and subsequently rating 4 sentences per scenario on how similar in meaning the (positive and negative) sentences are to the original scenario. Scores are based on how highly negative sentences are scored compared to positive sentences (i.e., higher scores = more negative interpretation bias).

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Given the small sample size and specific characteristics of the sample - there is increased likeliness of identifying someone who took part. Other researchers can request data - this will be reviewed by the team per request to ensure there is no possibility to identify any individuals.